CLINICAL TRIAL: NCT06049862
Title: "MaRiTensi" SELF MANAGEMENT APPLICATION FOR HYPERTENSION PATIENTS BASED ON M-HEALTH Its Effectiveness In Increasing Self- Care And Controlling Pressure Blood: Randomized Controlled Trial
Brief Title: The Effectiveness of "MaRiTensi" in Increasing Self-Care and Blood Pressure Control: Randomized Controlled Trial
Acronym: "MaRiTensi"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chatarina Setya Widyastuti (Other)
Collaborators: Gadjah Mada University (Other)
Responsible Party: Sponsor-Investigator, Chatarina Setya Widyastuti, S.Kep.,Ns.,M.Kep.,Sp.Kep.M.B, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KE/FK/0186/EC
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Primary Hypertension
Keywords: Hypertension; Mobile Health; Self-Management
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Intervention Model Description: The intervention was given in the third phase of the research, namely "MaRiTensi," which was developed in the first and second stages of the research.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: In the research, the third stage will do double-blinding for the care provider and outcome assessor, who will evaluate blood pressure and questionnaires. Allocation concealment for dividing into groups, intervention and control will use the SNOSE (sequentially numbered, opaque sealed envelopes ) method. The envelope closed will be sorted by order randomization, given paper carbon with appearance. The same is true for envelopes with the inscription intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MariTensi app and usual care (Experimental): Patients use the MaRitensi application to manage their hypertension by utilizing various menus in the application and continue receiving treatment as usual for 12 weeks.
  Interventions: Behavioral: MaRiTensi App
- Usual care (No Intervention): The patient was not given the MaRitensi application and only received treatment as usual.

INTERVENTIONS:
Behavioral: MaRiTensi App — MaRiTensi is a mobile health-based hypertension self-management application used on Android smartphones.
  MariTensi provides facilities for recording blood pressure, BMI, activity, examination results, education about hypertension, consultations, reminders and community chat.
  Arms: MariTensi app and usual care

SUMMARY:
This study aims to know the effectiveness of "MaRiTensi" in improving knowledge, motivation, efficacy, self-care and blood pressure control for hypertension patients.

This study hypothesizes that MaRiTensi effectively increases the knowledge, motivation, self-efficacy and self-care of hypertensive patients and reduces blood pressure in the intervention group compared to the control group.

Respondent recruitment is as follows:

1. The respondent candidate will be identified based on data on record medical
2. Appropriate respondent candidates' criteria inclusion and exclusion contacted for given informed consent
3. Prospective respondents who are willing to participate and fulfill the criteria for pressure blood moment measurement will request signed consent
4. Respondents fill in the basic data and recapitulate by the assistant researcher
5. Done randomization for allocation of group interventions and group control
6. Respondents given envelope closed (using sequentially numbered, opaque sealed envelopes (SNOSE) method )
7. Respondents' group intervention was given maintenance by Hospital or health center standard-added intervention using MaRiTensi by conditions; meanwhile, group control was provided care by Hospital or health center standards.

DETAILED DESCRIPTION:
Participants will be separated into two groups.

1. Respondents who have given consent will be given two questionnaires
2. Intervention group respondents will be given intervention for 12 weeks
3. Control group respondents will receive services according to the hospital or health center standards. Respondents will be asked to complete a questionnaire for the first evaluation during the first week of week six and to fill out a questionnaire for the final assessment in week 12.

Interventions in the form of utilizing "MaRiTensi" by the intervention group are given with the following conditions:

1. Intervention group and control group respondents filled out the Indonesian Version of the hypertension knowledge-level scale (HK-LS) questionnaire and the Indonesian Version of the Hypertension Self-care Profile (HBP-SCP)
2. Respondents were given a password to enter their data and log in to the "MaRiTensi" application.
3. Respondents will be given a simple and easy-to-understand tutorial on how to use "MaRiTensi."
4. Respondents measure blood pressure at least twice a week according to standards and record the results in the application
5. Respondents utilized every feature in MaRiTensi according to the needs of each respondent, including the question-and-answer feature
6. Respondents will be evaluated by telephone every two weeks by a research assistant to determine whether the respondent is following the intervention according to the procedure. Respondents who did not comply with the system were classified as lost follow-up
7. After using the "MaRiTensi" application, a post-test will be carried out at week six and week 12 using the Indonesian Version of the hypertension knowledge-level scale (HK-LS) and the Indonesian Version of the Hypertension Self-care Profile (HBP-SCP) questionnaire.

Data analysis in the third phase of the research was carried out by:

1. Editing Data originating from filling out the Indonesian Version of the hypertension knowledge scale (HK-LS) questionnaire and the Indonesian Version of the Hypertension Self-care Profile (HBP-SCP), as well as recording blood pressure in the application, will be examined for completeness, if there is incomplete data then will be asked back to the respondent to complete it.
2. Coding Coding will be provided for each questionnaire filled by respondents, especially for quantitative data according to the data scale. Coding is given according to the provisions in filling out the questionnaire (attached)
3. Tabulating Tabulating is done to convey respondents' demographic data in the third research and data on blood pressure, knowledge, motivation, self-efficacy, and self-care of hypertensive patients, as well as the results of the effectiveness analysis of "MaRiTensi" on these variables.

The data will be analyzed statistically using the paired t-test to analyze the first and second pre-test and post-test results. Comparison between the intervention and control groups will be analyzed by independent t-test. The first and second post-test outcome data will be subjected to an ANOVA test. All databases will be stored by researchers and validated by assessors, managed in a folder with a password so that not all teams can open it. Data analysis was carried out by the analyst, who performed it in a hidden manner, and the researcher will accept the data processing results for analysis to continue.

ELIGIBILITY:
Inclusion Criteria:

A patient registered in the medical record of RSPR, the doctor diagnosed with hypertension based on ICD 10: I10; Age 18 to <60 years; owning and being able to use a smartphone; living in Yogyakarta during the study period; blood pressure ≥ 140/90 mmHg measured at the time of visit.

Exclusion Criteria:

According to the doctor's diagnosis based on ICD 10:

1. Renal failure (ICD: N17-N19)
2. Diabetes Mellitus (ICD: E10-E14.9)
3. Stroke (ICD: I60-I69.8)
4. Acute Miocard Infarction (AMI) (ICD: I21-I21.9)
5. Heart Failure (ICD: I50-I50.9)
6. Cancer (ICD: C00-C97)
7. Dementia (ICD: F00-F04)
8. Mental disorders (ICD: F05-F99.9)
9. Thyroid Disease (ICD: E00-E07.9)
10. Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS) (ICD: B20)
11. Movement limitations: Hernia Nucleus Pulposus (HNP) (ICD: M50-M51.9); Piriformis Syndrome (ICD: G57-G57.9); Low Back Pain (LBP) (ICD: M54-M54.9); Frozen Shoulder (ICD: M75-75.9)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
The level of knowledge of hypertensive patients about hypertension | up to 12 weeks
  Everything that hypertensive patients know about, definitions, medical drugs, drug adherence, lifestyle, diet, and complications as measured by 22 questions using the Indonesian version of the HK-LS questionnaire
The motivation of hypertensive patients | up to 12 weeks
  The desire of hypertensive patients to take action to manage their hypertension as measured by 20 questions using the Indonesian version of the HBP-SCP questionnaire
Self-efficacy of hypertensive patients | up to 12 weeks
  A hypertensive patient's belief that he can manage his hypertension well as measured by 20 questions using the Indonesian version of the HBP-SCP questionnaire
Self-care of hypertensive patients | up to 12 weeks
  Actions initiated and performed by hypertensive patients to manage their disease as measured by 20 questions about self-management of hypertensive patients using the Indonesian version of the HBP-SCP questionnaire
Blood Pressure Control | up to 12 weeks
  A condition in which hypertensive patients can control their blood pressure. The criterion that blood pressure is under control if it meets 1 of the following criteria:
  1. There were no additional antihypertensive drugs during the study period
  2. There were no additional doses of antihypertensive drugs during the study period
  3. Blood pressure <140 mmHg at the first and second evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Chatarina S Widyastuti, Study Chair — Gadjah Mada University
Locations (3):
- Indonesia (3):
  - Puskesmas Depok 2, Sleman, D.I Yogyakarta
  - Puskesmas Pakem, Sleman, DI Yogyakarta
  - Panti Rapih Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: Yes
Data share to other reseacher for data analysis because there is a mask in data analysis in this study
Supporting Information: SAP
Time Frame: during study period
Access Criteria: numeric data for data analysis

REFERENCES:
- [Derived] Widyastuti CS, Dinarti LK, Aulawi K, Lazuardi L. Effectiveness of mHealth on self-care profile and blood pressure among patients with hypertension in Indonesia: A single-blind randomized controlled trial. Belitung Nurs J. 2025 May 27;11(3):294-304. doi: 10.33546/bnj.3760. eCollection 2025. PMID 40438651